CLINICAL TRIAL: NCT04842409
Title: Cardiological Monitoring and Safety of Ultra-hypofractionated Whole Breast Irradiation After Breast-conserving Surgery for Patients Affected by Breast Cancer: an Observational Prospective Cohort Study
Brief Title: Safety of Ultra-hypofractionated Whole Breast Irradiation After Breast-conserving Surgery
Acronym: SAFE-FORWARD
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Icro Meattini, M.D., Associate Professor, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: SAFE-FORWARD
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Radiotherapy Side Effect
Keywords: Breast Cancer; Radiotherapy; Safety
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Whole breast irradiation — Whole breast irradiation using an ultra-hypofractionated schedule (26 Gy in 5 fractions)

SUMMARY:
SAFE-FORWARD is an observational prospective cohort study. Patient population included both invasive and ductal carcinoma in situ (DCIS) breast cancer receiving ultra-hypofractionated whole breast irradiation (26 Gy in 5 fractions) after breast conserving surgery, as per physician choice. Adjuvant endocrine therapy as per local policy is allowed. Main exclusion criteria are mastectomy with or without breast reconstruction, neoadjuvant and/or adjuvant chemotherapy, and needs for a tumor bed radiation boost.

All enrolled patients will be prospectively monitored for 12 months, receiving a complex cardiological assessment before radiation therapy (RT) start (baseline), and at 2-, 6-, and 12-month after RT end of treatment. Both acute- , defined as adverse events recorded within the first 90 days since RT start, and early-late toxicity, will be scored according to EORTC (European Organisation for Research and Treatment of Cancer)/Radiation Therapy Oncology Group (RTOG) and CTCAE (v.5) scales.

Patients will undergo six-monthly follow-up clinical visits for the first 5 years and annual follow-up visits thereafter up to 10 year, as per clinical local practice. Breast cosmesis will be evaluated through the use of BCCT.core tool and assessment of the health-related quality of life will be performed through the EORTC quality of life questionnaire (QLQ) C30 and BR45 modules questionnaires at baseline, at the end of RT treatment, at 2- and 6-month.

DETAILED DESCRIPTION:
This prospective cohort study aims to assess heart toxicity and safety using a 1-week radiation schedule regimen of 26 Gy in five daily fractions.

The primary endpoint was defined as detection of any subclinical impairment in myocardial function and deformation (decrease ≥10%) measured with standard and 3-dimensional (3D) echocardiography and left ventricular (LV) global longitudinal strain (GLS).

Cardiac assessment. Medical history, electrocardiogram (EKG), clinical examination with specific attention to signs of heart failure, New York Heart Association (NYHA) class and Canadian angina grading scale score were recorded during each visit. Transthoracic echocardiography was performed with a commercially available system (EPIQ, X5-1 transducer, Philips Healthcare, Andover, Massachusetts). All measurements were performed and reported accordingly to the American Society of Echocardiography (ASE) and the European Association of Cardiovascular Imaging (EACVI) recommendations. Each measure was averaged over three cardiac cycles. Two-dimensional LVEF (2D-LVEF) was measured by Simpson rule, throughout apical 4- and 2-chamber views. LV mass was calculated from LV oriented M-mode tracings using the Devereux formula, ASE convention, and was indexed to body surface area (BSA). Diastolic function was evaluated by left atrial volume index, systolic pulmonary pressure, mitral inflow E/A pattern, E/A ratio, E velocity deceleration time, annular tissue Doppler e', and E/e' ratio. After optimizing image quality, maximizing frame rate, and minimizing foreshortening, which are all critical to reduce measurement variability, GLS measurements were made in the three standard apical views and averaged. LV 4-, 3-, and 2-chamber views were acquired during breath hold. From apical long-axis view to visualize aortic valve closure, using opening and closing clicks of the aortic valve the timing of aortic valve opening and closing on continuous wave (CW) Doppler imaging respect to EKG R wave was measured. Full-volume six-cycles gated acquisition breath hold images of left ventricle were acquired for Q-lab analysis to obtain end-diastolic volume, end systolic volume, indexed to BSA (EDVI and ESVI) and 3D-LVEF. Q-lab version in this study was 10.5. All echocardiography data was stored including the original Digital Imaging and Communications in Medicine (DICOM) images. All scans were read jointly by two experienced board certified echocardiographers who were blinded to all clinical characteristics. Systemic arterial pressure was measured simultaneously with echo measurements, by means of an arm-cuff sphygmomanometer.

ELIGIBILITY:
Inclusion Criteria:

* Invasive and ductal carcinoma in situ (DCIS) breast cancer
* Indication to ultra-hypofractionated whole breast irradiation
* Written informed consent
* Aged more than 18 years old

Exclusion Criteria:

* Neoadjuvant and adjuvant chemotherapy
* Tumor bed radiation boost prescription

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by both invasive and ductal carcinoma in situ (DCIS) breast cancer receiving ultra-hypofractionated whole breast irradiation (26 Gy in 5 fractions) after breast conserving surgery, as per physician choice. Adjuvant endocrine therapy as per local policy was allowed. Main exclusion criteria were mastectomy with or without breast reconstruction, neoadjuvant and/or adjuvant chemotherapy, and needs for a tumor bed radiation boost.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline 3-dimensional left ventricular ejection fraction (3D-LVEF) at 12 months | Baseline to 12-month
  Assessment of 3D-LVEF
Change from baseline Global Longitudinal Strain (GLS) at 12 months | Baseline to 12-month
  Assessment of GLS

CONTACTS AND LOCATIONS:
Overall Officials: Icro Meattini, MD, Prof, Principal Investigator — AOU Careggi; Lorenzo Livi, MD, Prof, Principal Investigator — AOU Careggi
Locations (1):
- Azienda Ospedaliero-Universitaria Careggi, Florence University, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided